CLINICAL TRIAL: NCT00350012
Title: Spatial Neglect and Bias in Near and Far Space
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, A. M. Barrett, MD, Director, Stroke Research, Kessler Foundation
Other Study IDs: K02NS047009; 5K02NS047099 (NIH)
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Stroke
Keywords: stroke; visual; spatial neglect
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Persons who have had a stroke and either have, or do not have, a pathological asymmetry of perception, attention and action causing functional disability (spatial neglect; Barrett and Burkholder, 2006).
- 2: Healthy age- and education-matched volunteers

SUMMARY:
The purpose of this research study is to learn how people distribute their visual attention when looking at objects nearby versus far away, and why vision may become distracted at near versus far distances.

DETAILED DESCRIPTION:
Visual distraction is a problem that more often occurs people who have suffered strokes than in the general population. Problems of visual attention generally appear immediately following a stroke, and may impair driving and other functions. While it is thought that there is a natural course of improvement over time, little is known about how this improvement occurs. Some studies suggest that recovery is only partial, meaning certain aspects of visual attention may improve while other aspects remain but escape notice.

The purpose of this study is to examine the effect of stroke on a person's visual attention when looking at objects nearby versus far away, and to learn why a person's visual attention may become more distracted at near versus far distances. The purpose of this study is also to understand how modeled interventions, such as eye patching or prism goggles, affect impairment measures of visual attention.

After an initial screening (including attention, thinking, memory, and visual judgment tests), participants will be given a neurological examination. Participants may be asked to perform visual tasks while wearing an eye patch or prism goggles. Next, they will be asked to perform a line bisection task by looking at lines on a video screen either at close or far distances and, using a laser pointer, marking the center of the lines as they appear on-screen. Participants may be asked to perform other, similar visual tasks as well.

Duration of the study for participants varies, ranging from 1 or 2 sessions totaling approximately 2 hours to multiple sessions spanning a year.

Research from this study may help researchers better understand problems associated with stroke and may lead to therapies designed to promote improved visual attention.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a history of stroke.
* The subject is 18 to 100 years old.
* The subject is able to give Informed consent.
* The subject is post-Stroke with left-hemisphere injury and has no spatial neglect (no attentional imbalance).
* The subject is post-stroke with right hemisphere damage and has spatial neglect (attentional imbalance).
* Healthy subject with no brain injury.
* The subject is post stroke and has hemianopia (a "visual field cut").
* The subject is able and willing to comply with the study protocol, including availability for all scheduled clinic visits.

Exclusion Criteria:

* Subjects with brain tumors, head injury with loss of consciousness, visual disorders other than corrected near or far-sightedness, history of learning disabilities, dementia or Alzheimer's Disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons who have had a stroke. Also, healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2004-05; Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Kessler Foundation Neglect Assessment Process | From 1 or 2 sessions totaling approximately 2 hours to multiple sessions in one year
  a performance based and behavioral measure for spatial neglect that utilizes and standardizes the administration of the Catherine Bergego Scale (CBS)

SECONDARY OUTCOMES:
Behavior Inattention Test Behavior Inattention Test | 2 weeks
  Conventional subtest, a set of paper and pencil test for spatial neglect
Barthel Index | 2 weeks
  A functional independence assessment of daily tasks

CONTACTS AND LOCATIONS:
Overall Officials: A. M. Barrett, MD, Principal Investigator — Stroke Rehabilitation Research, Kessler Foundation Research Center
Locations (1):
- Kessler Foundation, 1199 Pleasant Valley Way, West Orange, New Jersey, United States

REFERENCES:
- [Derived] Boukrina O, Chen P, Budinoska T, Barrett AM. Exploratory examination of lexical and neuroanatomic correlates of neglect dyslexia. Neuropsychology. 2020 May;34(4):404-419. doi: 10.1037/neu0000619. Epub 2020 Jan 30. PMID 31999167
- [Derived] Caulfield MD, Chen P, Barry MM, Barrett AM. Which perseverative behaviors are symptoms of spatial neglect? Brain Cogn. 2017 Apr;113:93-101. doi: 10.1016/j.bandc.2016.11.002. Epub 2017 Feb 3. PMID 28167411